CLINICAL TRIAL: NCT05594576
Title: Comparison of the ENDOCUFF VISION® Endoscopy Cap Coupled With GI GENIUS™ Artificial Intelligence Compared to Each Device Alone in Improving Colonic Adenoma Detection Rate During Colonoscopy
Acronym: COLODETECT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NIMAO/2021-2/LC-01
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Adenoma; Intestinal Polyps
Keywords: colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma; Intestinal Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ENDOCUFF VISION® Endoscopic Cap coupled with GI GENIUS™ Artificial Intelligence (AI) (Experimental)
  Interventions: Procedure: GI GENIUS™ artificial intelligence system; Procedure: ENDOCUFF VISION® endoscopic cap
- GI GENIUS™ Artificial Intelligence (AI) alone (Active Comparator)
- ENDOCUFF VISION® endoscopic cap alone (Active Comparator)
  Interventions: Procedure: ENDOCUFF VISION® endoscopic cap

INTERVENTIONS:
Procedure: GI GENIUS™ artificial intelligence system — Device used during coloscopy for detection of colonic adenoma
  Arms: ENDOCUFF VISION® Endoscopic Cap coupled with GI GENIUS™ Artificial Intelligence (AI)
Procedure: ENDOCUFF VISION® endoscopic cap — Device used during coloscopy for detection of colonic adenoma
  Arms: ENDOCUFF VISION® Endoscopic Cap coupled with GI GENIUS™ Artificial Intelligence (AI); ENDOCUFF VISION® endoscopic cap alone

SUMMARY:
Colorectal cancer is the 2nd most common cause of death by cancer. Screening is therefore essential, with a positive impact for prevention, and in the visualization and removal of colonic adenomas, pre-cancerous lesions of colorectal cancer.

The colonic adenoma detection rate (CADR), the gold standard for colonoscopy screening and screening studies, is the ratio of the number of colonoscopies with at least one histologically verified colonic adenoma to the total number of colonoscopies performed in a center. It varies between 25 and 45% depending on the center. There is a large inter-operator CADR variability, which has been linked to an increased incidence and excess mortality in colorectal cancers.

To improve this detection rate, several innovative techniques have been developed:

The endoscopic cap helps improve this detection rate: it is a 2cm tip with double row of plastic wings, fixed to the distal end of the colonoscope, which acts by unfolding the colonic haustrations allowing a better visualization of adenomas, and more particularly those of sessile morphology and sigmoidal location. Several multicenter studies have shown an improvement in the adenoma detection rate with this device compared to screening colonoscopy alone, with an adenoma detection rate optimization of 14%. Since then other devices, such as the Endocuff, have emerged with comparable efficacy. The Medtronic© GI GENIUS system integrates artificial intelligence (AI) to assist in the detection of polyps. It automatically identifies these precancerous lesions in real time.

The study investigators previously performed a retrospective pilot study (COLODETECT), comparing colonoscopy alone as a control group, against AI alone and against the combined cap + AI. This study showed encouraging results in terms of colonic adenoma detection rate (60% for the AI + cap group versus 37% for the AI alone group versus 33% for the colonoscopy alone group, p=0.037) However, it requires a higher level of evidence to be validated in practice. This prospective COLODETECT2 study estimated an a priori expected difference between A.I. - Cap and A.I. alone of about 15% CADR.

The GI GENIUS artificial intelligence system and the ENDOCUFF VISION endoscopic cap have separately proven their effectiveness in terms of colonic adenoma detection compared to colonoscopy alone. However, some limitations remain: existence of false positives (mucosal folds, residues), some morphological types still difficult to recognize (scalloped adenomas), non visualized colonic lesions.

This study therefore focuses on the possible complementarity of these 2 medical devices, in order to maximize the detection rate of colonic adenomas, and thus overcome the limitations of these two techniques by optimizing the visualization of these precancerous lesions, and consequently increasing the impact of colorectal cancer screening.

The study authors hypothesize that the combination of GI GENIUS™ AI coupled with the ENDOCUFF VISION® endoscopy cap provides a better colonic adenoma detection rate (CAD) during colonoscopy than either GI GENIUS™ AI alone or the ENDOCUFF VISION® cap alone.

ELIGIBILITY:
Inclusion Criteria:

* Need to perform colorectal cancer screening colonoscopy:

  * Primary Screening: Fecal Immunological Test positive;
  * Secondary screening: personal or family history of polyps, personal or family history of colorectal cancer, rectorrhagia-like symptomatology.
* Patient candidate for outpatient management.
* Patient who has given free and informed consent.
* Patient who has signed the consent form.
* Patient affiliated or beneficiary of a health insurance plan.

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* History of inflammatory bowel disease, Crohn's disease.
* Failure of a previous colonoscopy.
* Known familial polyposis.
* Contraindication to polypectomy (coagulation disorder, treatment with CLOPIDOGREL / anticoagulant).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Compare colonic adenoma detection rates (CADR) during colonoscopy between the three groups | Day 0
  %; defined as the number of colonoscopies with detection of at least one colonic adenoma out of the total number of colonoscopies performed

SECONDARY OUTCOMES:
Operator effect on CADR, between the three groups, per operator | Day 0
  CADR (%), defined as the number of colonoscopies with detection of at least one colonic adenoma out of the total number of colonoscopies performed for each strategy per operator
CADR according to adenoma size, for each strategy | Day 0
  CADR (%), detected by colonoscopy according to their size in mm (especially those smaller than 3 mm)
CADR according to adenoma histology for each strategy. | Day 0
  CADR (%), detected by colonoscopy according to histology (low/high grade dysplasia)
CADR according to adenoma morphology for each strategy. | Day 0
  CADR (%), detected by colonoscopy according to (Paris morphological classification: Ip, Is, IIa, IIb, IIc, III)
Shrinkage time for the Genius groups. | Day 0
  Measurement of withdrawal time (min, sec) for GI GENIUS™-Cap software or GI GENIUS™ software alone strategies (time from cecum to colonoscope removal).
Rate of cecal intubation between groups | Day 0
  % of exams in which the entire colon was examined.
Progression time between groups | Day 0
  Mean progression time (time from introduction of colonoscope to cecum; min, sec
Operative time between groups | Day 0
  Mean time from introduction of colonoscope to removal of endoscope from patient; min, sec
The number of immediate intra- and postoperative adverse events (bleeding, perforation) according to the different strategies | Day 0
  Collection of immediate intra- and postoperative adverse events (bleeding, perforation) for the three study strategies

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic Caillo, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - CHU de Limoges, Limoges
  - CHU de Nîmes, Nîmes